CLINICAL TRIAL: NCT06787547
Title: A Prospective, Multi-center, Single-arm, Objective Performance Goal Pre-specified Study to Evaluate the Safety and Effectiveness of Intravascular Lithotripsy Generator Combined with SONICO-CX Coronary Intravascular Lithotripsy (IVL) Catheter for Pre-treatment of Coronary Calcification Before Stent Implantation
Brief Title: Effectiveness and Safety of a Novel Intravascular Lithotripsy System in Severely Calcified Coronary Lesions(COCALP)
Acronym: COCALP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectrumedics Medical Technology(Shanghai)Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-120R
Record Dates: First submitted 2025-01-14; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Calcified Coronary Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Patients underwent Intravascular lithotripsy (IVL) (Experimental): Patients with severely calcified coronary lesions were enrolled and underwent IVL
  Interventions: Device: IVL(Sonico-CX)

INTERVENTIONS:
Device: IVL(Sonico-CX) — SONICO-CX® balloon matched 1:1 to the reference vessel diameter, was advanced to the target lesion to pretreat

SUMMARY:
This study is a prospective, multicenter, single-arm trial designed to investigate the effectiveness and safety of this intravascular lithotripsy system to treat severely calcified coronary lesions before stenting.

DETAILED DESCRIPTION:
Subject Population: Subjects ≥ 18 years of age with de novo, calcified coronary artery lesions presenting with stable, unstable or silent ischemia that are suitable for percutaneous coronary intervention (PCI). 266 subjects at 11 sites will be enrolled.Subjects will be followed through discharge, 30 days, 6months.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria

  1. Age ≥ 18 years old
  2. Evidence of asymptomatic ischemia, stable or unstable angina
  3. Patients who can understand the purpose of the trial, voluntarily participate and sign informed consent, and are willing to undergo angiography, OCT, and clinical follow-up.
* Angiographic Inclusion Criteria

  1. The target lesion must be a de novo coronary lesion that has not been previously treated with any interventional procedure
  2. Length of the target lesion ≤60mm, diameter of the target lesion 2.5-4.0mm
  3. Target lesion diameter stenosis ≥70%, the doctor determines the need for stent implantation
  4. The lesion allows 0.014 guide wires to pass through
  5. Under multi-angle contrast conditions, it can be seen that there are calcified angiography lesions on both sides of the lesion blood vessel wall (the target lesion meets the definition of severe calcification).

Exclusion Criteria:

* General inclusion criteria

Patients who fit any of the following criteria were excluded:

1. Acute myocardial infarction occurred within 30 days before procedural
2. Simultaneous use of spinning or special balloons (chocolate balloons, scoring balloons, spinous balloons, etc.) to treat the lesion
3. Troponin was 5 times greater than the upper limit of laboratory normal within one week before procedural
4. Severe cardiac insufficiency (Grade III or IV)
5. Left ventricular ejection fraction < 40%
6. The patient refuses emergency CABG surgery or does not have indications for emergency CABG surgery.
7. Uncontrolled severe hypertension (ystolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg)
8. Severe renal failure (serum creatinine > 221μmol/L)
9. Preprocedural hemoglobin < 100g/L
10. Significant coagulation dysfunction (platelet count < 100×109/L or INR>1.7, INR is only required for patients who have taken warfarin orally within 2 weeks prior to enrollment)
11. Hypercoagulable blood disorders (e.g. Polycythemia vera, platelet count >750× 109/L, etc.)
12. History of stroke or TIA within 3 months
13. History of active digestive ulcer or upper gastrointestinal bleeding within 6 months
14. The patients has a life expectancy of less than 12 months
15. The patient has an active systemic infection
16. The patient has a connective tissue disease (such as Marfan's syndrome)
17. The patient is allergic to contrast material
18. Patients undergoing heart transplantation
19. Patients with pacemakers implanted
20. The patient is pregnant or breastfeeding
21. Those who have participated in clinical trials of other drugs or medical devices within 1 month before enrollment
22. Other circumstances that the investigator deems inappropriate to participate in the trial - Angiographic Exclusion Criteria

Patients who met any of the following criteria were excluded:

1. Unprotected left main disease (left main visual stenosis > 50%)
2. Baseline TIMI blood flow less than grade 3 (allows evaluation after pre-dilation)
3. A stent has been implanted within 10mm of the proximal or distal end of the target lesion
4. The target lesion is located at the distal end of the saphenous vein or LIMA/RIMA bypass graft
5. Aneurysm within the target blood vessel
6. Angiography confirmed the presence of thrombus in the target vessel
7. Chronic total occlusive lesions
8. Angiography confirmed the presence of severe dissection of the target lesion prior to hydroelectric shock wave lithotripsy treatment (D-F dissection (NHLBI classification)）
9. The investigators determined that the target lesion was unsuitable for patients undergoing vasodilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Procedural success rate | During hospitalization (up to 7 days after operation)
  defined as successful stent implantation with ≤30% in-stent residual stenosis and the absence of in-hospital MACE, including cardiac death, MI, and target vessel revascularization

SECONDARY OUTCOMES:
Angiography success rate | Immediately after operation
  Angiographic success was defined as successful stent implantation with ≤30% in-stent residual stenosis and without serious angiographic complications immediately after IVL, including type D to F severe dissection, perforation, acute occlusion, sustained slow-flow, or no-reflow
Device success rate | Immediately after operation
  Device success was defined as the IVL catheter successfully crossing the target lesion and delivering lithotripsy without serious angiographic complications immediately following the procedure
MACE events | before discharge, 30 days and 6 months post-procedural
  MACE--a composite of cardiac death, myocardial infarction (MI) and target vessel revascularization (TVR)

OTHER OUTCOMES:
Adverse Events | before discharge, 30 days and 6 months post-procedural
  Incidence of other adverse events during procedural, before discharge, 30 days and 6 months post-procedural

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - First Affiliated Hospital of University of Science and Technology of China,, Hefei, Anhui
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tongji Hospital, Tongji University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Ningbo First Hospital University, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No